CLINICAL TRIAL: NCT06955572
Title: Descriptive Study of the Gene Count in Faecal Microbiota During the Course of Various Pathologies and Correlation With the Clinical Phenotype
Brief Title: Descriptive Study of the Gene Count in Faecal Microbiota
Acronym: METARICH
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/196/OB; ID RCB : 2022-A01921-42 (Other: ANSM)
Record Dates: First submitted 2025-04-24; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Microbiota
Keywords: faecal microbiota
MeSH Terms: interventions — Adiposity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human faeces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients with colorectal cancer — Analysis of the lower fecal gene count (fGC) compared with the control group
Diagnostic Test: Patients with Parkinson's disease — Analysis of the lower fecal gene count (fGC) compared with the control group
Diagnostic Test: Patients with non-alcoholic steatohepatitis — Analysis of the lower fecal gene count (fGC) compared with the control group
Diagnostic Test: Patients with obesity — Analysis of the lower fecal gene count (fGC) compared with the control group
Diagnostic Test: Healthy volunteers — Determination of the number of bacterial faecal genes (fGC, fecal Gene Count) inferior reference

SUMMARY:
The hypothesis of METARICH Study is that it is possible to draw up a profile of the faecal microbiota, which could contribute in the future to the characterisation of certain chronic pathologies. The pathologies chosen for the study were selected because they are associated in the literature with changes in the faecal microbiota.

DETAILED DESCRIPTION:
All the study data will be collected from the patients' clinical records and from the questionnaires set up (patient inclusion questionnaire and information questionnaire).

* The patient inclusion questionnaires collect the following variables: characteristics of the pathology (precise phenotyping by the clinician, assessment of severity, age, progression) as well as biological parameters obtained in the patient's usual check-ups and current treatments specific to the pathology.
* The patient information questionnaire collects information on lifestyle habits (smoking, alcohol, sporting activities, diet), stool sample data (Bristol scale, day and time of collection), treatment(s) received in the last 3 months and other chronic pathologies.

ELIGIBILITY:
Inclusion Criteria:

List of patient inclusion criteria:

Male or female patient consulting the Rouen University Hospital for one of the 4 pathologies below:

* Obesity (with or without bulimic hyperphagia): BMI greater than 30
* Non-alcoholic steatohepatitis (NASH): Confirmation of the diagnosis of NASH by the clinician
* Colorectal cancer: Confirmation of the diagnosis of colorectal cancer by the clinician
* Parkinson's disease: Confirmation of the diagnosis of Parkinson's disease by the clinician

List of inclusion criteria for the control group:

* Adult patient aged less than 75 years.
* Ambulatory patient able to collect stools at home
* Patient who has read and understood the information letter and signed the consent form
* Patient affiliated to the social security system
* Aged between 18 and 75
* Affiliated with a social security scheme
* To the best of the volunteer's knowledge, free from the following pathologies: Obesity, hyperphagia, anorexia, bulimia, Crohn's disease, irritable bowel syndrome, haemorrhagic rectocolitis, NASH, steatosis, colorectal cancer, diabetes (type I and II), ankylosing spondylitis, rheumatoid arthritis, heart failure, atopic dermatitis, bronchopulmonary concer, Parkinson's disease and multiple sclerosis
* A person who has read and understood the information leaflet, signed the consent forms and is able to perform the stool collection.

Exclusion Criteria:

List of patient non-inclusion criteria :

* Patient under guardianship or incapable of giving consent
* Patient at the end of life or whose clinical condition is incompatible with stool collection
* Patient undergoing antibiotic therapy or who has received antibiotic therapy for less than 3 months
* Patient already included in a category 1 interventional clinical trial
* Patient already included in METARICH for another pathology
* Patient who has had a colonic lavage/emptying for less than 3 months

List of non-inclusion criteria for the control group:

* Person deprived of liberty by administrative or judicial decision or person subject to a legal adult protection measure, patient under court protection, patient under guardianship or curatorship,
* Person under antibiotic therapy or having received antibiotic therapy for less than 3 months
* Person already included in a category 1 interventional clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 patients with non-alcoholic steatohepatitis, 60 patients with colorectal cancer, 60 patients with Parkinson's disease, 80 patients 60 patients with obesity and 140 healthy volunteers will be selected.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Gene richness of faecal microbiota | At enrollment visit, Month 2
  Measuring the gene richness of faecal microbiota in Patients with colorectal cancer arm
Gene richness of faecal microbiota | At enrollment visit, Month 2
  Measuring the gene richness of faecal microbiota in Patients with obesity arm
Gene richness of faecal microbiota | At enrollment visit, Month 2
  Measuring the gene richness of faecal microbiota in Patients with Parkinson's disease arm
Gene richness of faecal microbiota | At enrollment visit, Month 2
  Measuring the gene richness of faecal microbiota in Patients with non-alcoholic steatohepatitis arm
Gene richness of faecal microbiota | At enrollment visit, Month 2
  Measuring the gene richness of faecal microbiota in Healthy volunteers arm

SECONDARY OUTCOMES:
Diversity of bacterial species | At enrollment visit, Month 2
  Gene counting from metagenomic sequencing in Patients with colorectal cancer arm
Diversity of bacterial species | At enrollment visit, Month 2
  Gene counting from metagenomic sequencing in Patients with obesity arm
Diversity of bacterial species | At enrollment visit, Month 2
  Gene counting from metagenomic sequencing in Patients with Parkinson's disease arm
Diversity of bacterial species | At enrollment visit, Month 2
  Gene counting from metagenomic sequencing in Patients with non-alcoholic steatohepatitis arm
Diversity of bacterial species | At enrollment visit, Month 2
  Gene counting from metagenomic sequencing in Healthy volunteers arm
Metagenomic data library | At enrollment visit, Month 2
  Creation of a metagenomic data library referencing the data collected
Discriminating gene count threshold | At enrollment visit, Month 2
  Identify a gene count threshold that discriminates against the degree of severity of the disease (colorectal cancer)
Discriminating gene count threshold | At enrollment visit, Month 2
  Identify a gene count threshold that discriminates against the degree of severity of the disease (obesity)
Discriminating gene count threshold | At enrollment visit, Month 2
  Identify a gene count threshold that discriminates against the degree of severity of the disease (Parkinson)
Discriminating gene count threshold | At enrollment visit, Month 2
  Identify a gene count threshold that discriminates against the degree of severity of the disease (non-alcoholic steatohepatitis)

CONTACTS AND LOCATIONS:
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.